CLINICAL TRIAL: NCT06561386
Title: A Phase 3, Randomized, Open-label Study of Nivolumab + Relatlimab Fixed-dose Combination With Chemotherapy Versus Pembrolizumab With Chemotherapy as First-line Treatment for Participants With Non-squamous (NSQ), Stage IV or Recurrent Non-small Cell Lung Cancer and With Tumor Cell PD-L1 Expression ≥ 1%
Brief Title: A Study to Compare the Efficacy of Nivolumab and Relatlimab Plus Chemotherapy vs Pembrolizumab Plus Chemotherapy for Stage IV/Recurrent Non-squamous Non-small Cell Lung Cancer With PD-L1 Expression ≥ 1%
Acronym: RELATIVITY1093
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA224-1093; 2024-513682-40 (Other: EU CTR); U1111-1306-8896 (Other: WHO)
Record Dates: First submitted 2024-08-16; First posted 2024-08-20 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-squamous; PDL-1 ≥ 1%
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab; relatlimab; pembrolizumab; Carboplatin; Pemetrexed; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental)
  Interventions: Drug: Nivolumab; Drug: Relatlimab; Drug: Carboplatin; Drug: Pemetrexed; Drug: Cisplatin
- Arm B (Active Comparator)
  Interventions: Drug: Pembrolizumab; Drug: Carboplatin; Drug: Pemetrexed; Drug: Cisplatin

INTERVENTIONS:
Drug: Nivolumab — Specified dose on specified days
  Arms: Arm A
Drug: Relatlimab — Specified dose on specified days
  Arms: Arm A
Drug: Pembrolizumab — Specified dose on specified days
  Arms: Arm B
Drug: Carboplatin — Specified dose on specified days
Drug: Pemetrexed — Specified dose on specified days
Drug: Cisplatin — Specified dose on specified days

SUMMARY:
The purpose of this study is to compare the efficacy of Nivolumab and Relatlimab in combination with chemotherapy to Pembrolizumab with Chemotherapy in participants with stage IV or recurrent Non-squamous Non-small Cell Lung Cancer with PD-L1 expression ≥ 1%

ELIGIBILITY:
Inclusion Criteria

* Participants must have histologically confirmed Stage IV or recurrent Non-small Cell Lung Cancer (NSCLC) of non-squamous (NSQ) histology with no prior systemic anti-cancer therapy given as primary therapy for advanced or metastatic disease.
* Participants must have measurable PD-L1 ≥ 1% Tumor Cell (TC) score by the investigational PD-L1 immunohistochemistry (IHC) assay VENTANA PD-L1 (SP263) CDx Assay conducted by central laboratory during the screening period prior to randomization.
* Participants must have measurable disease by computed tomography (CT) or magnetic resonance imaging (MRI) per RECIST v1.1 criteria.
* Participants must have an Easter Cooperative Oncology Group (ECOG) performance status of ≤ 1 at screening.
* Participants must have a life expectancy of at least 3 months at the time of randomization.

Exclusion Criteria

* Participants must not be pregnant and/or breastfeeding.
* Participants with epidermal growth factor receptor (EGFR), anaplastic lymphoma kinase (ALK), or ROS-1 mutations that are sensitive to available targeted inhibitor therapy. Participants with unknown EGFR, ALK, or ROS-1 status are excluded.
* Participants with known BRAFV600E mutations, that are sensitive to available targeted inhibitor therapy; participants with known activating rearranged during transfection (RET) mutations or neurotrophic tyrosine receptor kinase (NTRK) fusion gene alterations are excluded. Participants with unknown or indeterminate BRAF mutation, activating RET mutations or NTRK fusion gene alterations are eligible.
* Participants must not have untreated central nervous system (CNS) metastases.
* Participants must not have leptomeningeal metastases (carcinomatous meningitis).
* Participants must not have concurrent malignancy requiring treatment.
* Participants must not have an active autoimmune disease.
* Participants must not have history of interstitial lung disease or pneumonitis that required oral or intravenous (IV) glucocorticoids to assist with management.
* Participants must not have a history of myocarditis.
* Participants must not have had prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, or anti-CTLA-4 antibody, or other antibody or drug targeting T-cell co-stimulation or checkpoint pathways.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2024-10-07 (Actual); Primary Completion 2030-07-30 (Estimated); Study Completion 2032-08-04 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) in randomized participants with PD-L1 1% to 49% | Up to 5 years

SECONDARY OUTCOMES:
OS in randomized participants with PD-L1 ≥ 1% | Up to 5 years
Progression-free survival (PFS) as assessed by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) per blinded independent central review (BICR) | Up to 5 years
Overall response rate (ORR) | Up to 5 years
Duration of response (DoR) | Up to 5 years
Number of participants with adverse events (AEs) | Up to 2.5 years
Number of participants with serious adverse events (SAEs) | Up to 2.5 years
Number of participants with immune-mediated adverse events (IMAEs) | Up to 2.5 years
The time until definitive deterioration based on non-small cell lung cancer - symptom assessment questionnaire (NSCLC-SAQ) total score | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (278):
- United States (36):
  - Southern Arizona VA Health Care System, Tucson, Arizona
  - Local Institution - 0112, Los Angeles, California
  - University of California Davis (UC Davis) Comprehensive Cancer Center, Sacramento, California
  - San Francisco Oncology Associates, San Francisco, California
  - UCLA Hematology/Oncology - Santa Monica, Santa Monica, California
  - University of Miami Hospital and Clinics, Sylvester Cancer Center, Miami, Florida
  - Memorial Hospital West, Pembroke Pines, Florida
  - Florida Cancer Specialists - North, St. Petersburg, Florida
  - Florida Cancer Specialists - East, West Palm Beach, Florida
  - Affiliated Oncologists, LLC, Chicago Ridge, Illinois
  - Saint Elizabeth Medical Center Edgewood, Edgewood, Kentucky
  - Local Institution - 0130, Lexington, Kentucky
  - Hattiesburg Clinic Hematology/Oncology, Hattiesburg, Mississippi
  - Local Institution - 0308, Bozeman, Montana
  - Renown Regional Medical Center, Reno, Nevada
  - St. Joseph's Regional Medical Center, Paterson, New Jersey
  - New Mexico VA Healthcare System, Albuquerque, New Mexico
  - WMCHealth Advanced Physician Services, Hawthorne, New York
  - Veterans Affairs New York Harbor Healthcare System, New York, New York
  - Local Institution - 0380, Northport, New York
  - University of Rochester Medical Center, Rochester, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Local Institution - 0357, The Bronx, New York
  - Messino Cancer Centers, Asheville, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Local Institution - 0369, Canton, Ohio
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Louis Stokes Cleveland VA Medical Center, Cleveland, Ohio
  - Local Institution - 0366, Massillon, Ohio
  - Lancaster General Hospital - Ann B Barshinger Cancer Institute, Lancaster, Pennsylvania
  - Local Institution - 0464, Nashville, Tennessee
  - Texas Oncology - West Texas, Abilene, Texas
  - Local Institution - 0305, Harlingen, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - The University of Texas Health Science Center at Tyler dba UT Health East Texas HOPE Cancer Center, Tyler, Texas
  - Local Institution - 0302, Salt Lake City, Utah
- Argentina (8):
  - Hospital Británico de Buenos Aires, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Instituto Alexander Fleming, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Hospital Italiano de Buenos Aires, ABB, Buenos Aires F.D.
  - Instituto Médico Río Cuarto, Río Cuarto, Córdoba Province
  - Sanatorio Parque, Rosario, Santa Fe Province
  - Hospital Privado Universitario de Córdoba, Córdoba
  - Instituto Oncológico de Córdoba, Córdoba
  - Hospital Privado de Comunidad, Mar del Plata
- Australia (8):
  - Gosford Hospital, Gosford, New South Wales
  - GenesisCare North Shore, St Leonards, New South Wales
  - The Prince Charles Hospital, Brisbane, Queensland
  - Gallipoli Medical Research Ltd, Brisbane, Queensland
  - Local Institution - 0057, Elizabeth Vale, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - St. John of God Murdoch Hospital, Murdoch, Western Australia
- Austria (3):
  - Universitätsklinikum Krems, Krems, Lower Austria
  - Klinikum Wels-Grieskirchen GmbH, Wels, Upper Austria
  - Klinik Floridsdorf, Vienna
- Belgium (6):
  - Antwerp University Hospital, Edegem, Antwerpen
  - UZ Brussel, Brussels, Bruxelles-Capitale, Région de
  - Jessa Ziekenhuis, Hasselt, Limburg
  - Université Catholique de Louvain-Namur - Centre Hospitalier Universitaire Dinant-Godinne - Site Godinne, Yvoir, Namur
  - AZ Delta vzw, Roeselare, West-Vlaanderen
  - Centre Hospitalier Universitaire de Liège - Domaine Universitaire du Sart Tilman, Liège
- Brazil (12):
  - Pronutrir, Fortaleza, Ceará
  - Cetus Oncologia - Unidade Belo Horizonte, Belo Horizonte, Minas Gerais
  - CTO - Centro de Tratamento Oncológico, Belém, Pará
  - Liga Norte Riograndense Contra o Câncer, Natal, Rio Grande do Norte
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital São Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - Clínica de Neoplasias Litoral, Itajaí, Santa Catarina
  - Fundação Pio XII - Hospital de Câncer de Barretos, Barretos, São Paulo
  - NAIC - Instituto do Câncer, Bauru, São Paulo
  - Centro de Oncologia - CEON+ - Unidade São Caetano do Sul, São Caetano do Sul, São Paulo
  - Instituto Nacional de Câncer - INCA, Rio de Janeiro
  - Icesp - Instituto Do Câncer Do Estado de São Paulo, São Paulo
- Chile (5):
  - Oncocentro Apys, Viña del Mar, Región de Valparaíso
  - Orlandi Oncologia, Santiago, Santiago Metropolitan
  - Fundacion Arturo Lopez Perez (FALP), Santiago, Santiago Metropolitan
  - Pontificia Universidad Catolica de Chile, Santiago, Santiago Metropolitan
  - Bradfordhill, Santiago, Santiago Metropolitan
- China (31):
  - Local Institution - 0182, Hefei, Anhui
  - Beijing Cancer hospital, Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Chongqing Three Gorges Central Hospital, Wanzhou, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Huizhou Central People's Hospital, Huizhou, Guangdong
  - Liuzhou People's Hospital, Liuchow, Guangxi
  - Guangxi Medical University Affiliated Tumor Hospital, Nanning, Guangxi
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - The First Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan
  - Local Institution - 0237, Zhengzhou, Henan
  - Local Institution - 0235, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - First Huai'an Hospital Affiliated to Nanjing Medical University, Huai'an, Jiangsu
  - The First affiliated hospital of Nanchang University (Xianghu campus), Nanchang, Jiangxi
  - Liaoning Cancer Hospital, Shenyang, Liaoning
  - Xi'an International Medical Center Hospital, Xi'an, Shaanxi
  - Shandong Cancer Hospital, Jinan, Shandong
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Zhongshan Hospital,Fudan University, Shanghai, Shanghai Municipality
  - Shanxi Cancer Hospital, Taiyuan, Shanxi
  - Sichuan Cancer hospital, Chengdu, Sichuan
  - The Second People's Hospital of Neijiang, Neijiang, Sichuan
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - The first Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Linhai, Zhejiang
  - Guangdong Provincial People's Hospital, Guangzhou
- Colombia (6):
  - Local Institution - 0415, Medellín, Antioquia
  - Local Institution - 0443, Bogotá, Bogota D.C.
  - Local Institution - 0418, Bogotá, Bogota D.C.
  - Local Institution - 0417, Valledupar, Cesar Department
  - Local Institution - 0416, Pereira, Risaralda Department
  - Local Institution - 0442, Cali, Valle del Cauca Department
- Denmark (3):
  - Aarhus Universitetshospital, Skejby, Aarhus, Central Jutland
  - Sygehus Soenderjylland, Sønderborg, Region Syddanmark
  - Rigshospitalet, Copenhagen
- France (12):
  - CHRU de Brest, Brest, Finistère
  - CHU de Toulouse - Hopital Larrey, Toulouse, Haute-Garonne
  - Local Institution - 0092, Montpellier, Hérault
  - Local Institution - 0093, Rennes, Ille-et-Vilaine
  - Centre Hospitalier Régional Universitaire de Nancy - Hôpitaux de Brabois, Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - CHU Lille - Institut Coeur Poumon, Lille, Nord
  - Centre Hospitalier intercommunal de Toulon La Seyne sur Mer, Toulon, Provence-Alpes-Côte d'Azur Region
  - Centre Hospitalier Lyon Sud, Pierre-Bénite, Rhône
  - Centre Hospitalier de la Côte Basque, Bayonne
  - Assistance Publique Hôpitaux de Marseille - Hôpital Nord, Marseille
  - Hopitaux Universitaires Paris Centre-Hopital Cochin, Paris
  - Institut Curie, Paris
- Germany (14):
  - Klinikum Esslingen, Esslingen am Neckar, Baden-Wurttemberg
  - Bundeswehrkrankenhaus Ulm, Ulm, Baden-Wurttemberg
  - Local Institution - 0287, Kempten (Allgäu), Bavaria
  - Klinikum der Ludwig-Maximilians-Universitaet Muenchen, München, Bavaria
  - Universitätsklinikum Marburg, Marburg, Hesse
  - Praxis Onkologie am Raschplatz, Hanover, Lower Saxony
  - Evangelisches Krankenhaus Herne - Eickel, Herne, North Rhine-Westphalia
  - Universitätsklinikum Münster - Albert Schweitzer Campus, Münster, North Rhine-Westphalia
  - Klinikum Chemnitz, Chemnitz, Saxony
  - LungenClinic Grosshansdorf, Großhansdorf, Schleswig-Holstein
  - Charité Campus Virchow-Klinikum, Berlin
  - Universitätsklinikum Bonn, Bonn
  - Universitaetsklinikum Essen, Essen
  - Asklepios Klinik Gauting GmbH, Gauting
- India (9):
  - Local Institution - 0333, Bengaluru, Karnataka
  - Regional Cancer Centre - Thiruvananthapuram, Thiruvananthapuram, Kerala
  - Mumbai Oncocare Centre Vile Parle, Mumbai, Maharashtra
  - Tata Memorial Hospital, Mumbai, Maharashtra
  - All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi
  - Local Institution - 0448, New Delhi, National Capital Territory of Delhi
  - Rajiv Gandhi Cancer Institute And Research Centre, New Delhi, National Capital Territory of Delhi
  - Yashoda Hospital, Secunderabad, Telangana
  - Narayana Superspecialty Hospital, Howrah, West Bengal
- Ireland (4):
  - St. James's Hospital, Dublin
  - Local Institution - 0028, Dublin
  - Tallaght University Hospital, Dublin
  - Local Institution - 0027, Dublin
- Italy (9):
  - Instituto Tumori Giovanni Paolo II, Bari, Apulia
  - Ospedale Santa Maria delle Croci, Ravenna, Emilia-Romagna
  - Local Institution - 0045, Monza, Lombardy
  - Local Institution - 0465, Milan, Milano
  - A.O.R.N. Ospedale dei Colli - Monaldi V., Naples, Napoli
  - Local Institution - 0049, Naples, Napoli
  - Istituto Nazionale Tumori Regina Elena, Rome, Roma
  - Casa di Cura Dott. Pederzoli, Peschiera del Garda, Verona
  - Local Institution - 0222, Ravenna
- Japan (21):
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - University of Occupational and Enviromental Health, Kitakyushu, Fukuoka
  - Kurume University Hospital, Kurume, Fukuoka
  - Chugoku Central Hospital, Fukuyama-shi, Hiroshima
  - National Hospital Organization Hokkaido Cancer Center, Sapporo, Hokkaido
  - Kanagawa Cardiovascular and Respiratory Center, Yokohama, Kanagawa
  - Kanagawa cancer center, Yokohama, Kanagawa
  - Kochi Medical School Hospital, Nankoku, Kochi
  - Sendai Kousei Hospital, Sendai, Miyagi
  - Nara Medical University Hospital, Kashihara, Nara
  - Niigata Cancer Center Hospital, Niigata, Niigata
  - Kurashiki Central Hospital, Kurashiki, Okayama-ken
  - Kansai Medical University Hospital, Hirakata, Osaka
  - Kindai University Hospital, Sakai, Osaka
  - Saitama Medical University International Medical Center, Hidaka, Saitama
  - Hamamatsu University Hospital, Hamamatsu, Shizuoka
  - Shizuoka Cancer Center, Nagaizumi-cho,Sunto-gun, Shizuoka
  - The Cancer Institute Hospital of JFCR, Koto, Tokyo
  - Hyogo Cancer Center, Akashi
  - Fukushima Medical University, Fukushima
  - Osaka International Cancer Institute, Osaka
- Mexico (4):
  - Cancer Treamtent Clinic and Clinical Trials Sa de Cv, Guadalajara, Jalisco
  - Hospital H+ Queretaro, Querétaro City, Querétaro
  - Arké SMO S.A. de C.V., México
  - Centro Potosino de Investigación Médica, San Luis Potosí City
- Netherlands (8):
  - Local Institution - 0030, Harderwijk, Gelderland
  - Atrium-Orbis - Zuyderland Medisch Centrum Heerlen, Heerlen, Limburg
  - Local Institution - 0196, 's-Hertogenbosch, North Brabant
  - Local Institution - 0195, Zwolle, Overijssel
  - Leids Universitair Medisch Centrum, Leiden, South Holland
  - Local Institution - 0315, The Hague, South Holland
  - Ziekenhuis Rijnstate, Arnhem
  - Local Institution - 0032, Groningen
- New Zealand (5):
  - Local Institution - 0407, Tauranga, Bay of Plenty
  - Tauranga Hospital, Tauranga, Bay of Plenty
  - Auckland City Hospital, Auckland
  - Local Institution - 0425, Dunedin
  - Local Institution - 0406, Wellington
- Poland (8):
  - Local Institution - 0255, Konin, Greater Poland Voivodeship
  - Centrum Medyczne Pratia Poznań, Poznan, Greater Poland Voivodeship
  - Local Institution - 0261, Poznan, Greater Poland Voivodeship
  - Centrum Onkologii im. Prof. Franciszka Lukaszczyka, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Local Institution - 0259, Warsaw, Masovian Voivodeship
  - Local Institution - 0257, Koszalin, West Pomeranian Voivodeship
  - Szpital Specjalistyczny w Prabutach Spolka z o.o., Prabuty
  - Instytut Centrum Zdrowia Matki Polki, Lodz, Łódź Voivodeship
- Portugal (4):
  - Instituto Português de Oncologia de Lisboa Francisco Gentil, Lisbon, Lisbon District
  - Local Institution - 0404, Coimbra
  - Instituto Português de Oncologia do Porto Francisco Gentil, EPE, Porto
  - Local Institution - 0401, Porto
- Romania (7):
  - SC Memorial Healthcare International SRL, Bucharest, București
  - Institutul Oncologic Bucuresti "Prof. Dr. Alexandru Trestioreanu", Bucharest, București
  - SC Radiotherapy Center Cluj SRL, Florești, Cluj
  - Centrul de Oncologie "Sfântul Nectarie", Craiova, Dolj
  - Institutul Oncologic Cluj, Cluj-Napoca
  - Institutul Regional de Oncologie, Iași
  - Spitalul Municipal Schuller Ploiești, Ploieşti
- Saudi Arabia (3):
  - Local Institution - 0440, Dammam, Eastern Province
  - Local Institution - 0409, Jeddah, Makkah Al Mukarramah
  - Local Institution - 0408, Riyadh, Riyadh Region
- South Africa (5):
  - Local Institution - 0429, Johannesburg, GP
  - Local Institution - 0432, Pretoria, GP
  - Local Institution - 0427, Sandton, GP
  - Local Institution - 0431, Soweto, GP
  - Local Institution - 0428, Cape Town, Western Cape
- South Korea (9):
  - Chungbuk National University Hospital, Cheongju-si, Chungcheongbuk-do [Chungbuk]
  - Gachon University Gil Medical Center, Namdong-gu, Incheon-gwangyeoksi [Incheon]
  - Chonnam National University Hwasun Hospital, Hwasun, Jeonranamdo
  - National Cancer Center, Goyang-si, Kyǒnggi-do
  - CHA Bundang Medical Center, CHA University, Seongnam-si, Kyǒnggi-do
  - Pusan National University Hospital, Busan, Pusan-Kwangyǒkshi
  - Severance Hospital, Yonsei University Health System, Seoul, Seoul-teukbyeolsi [Seoul]
  - Asan Medical Center, Seoul, Seoul-teukbyeolsi [Seoul]
  - Samsung Medical Center, Seoul, Seoul-teukbyeolsi [Seoul]
- Spain (12):
  - CHUAC-Hospital Teresa Herrera, A Coruña, A Coruña [La Coruña]
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona [Barcelona]
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalunya [Cataluña]
  - Local Institution - 0267, L'Hospitalet de Llobregat, Catalunya [Cataluña]
  - Hospital Son Llàtzer, Palma, Illes Balears [Islas Baleares]
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid, Comunidad de
  - Hospital Universitario 12 de Octubre, Madrid, Madrid, Comunidad de
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid, Comunidad de
  - Local Institution - 0411, Valencia, València
  - H.R.U Málaga - Hospital General, Málaga
  - Hospital Universitario Virgen Del Rocio, Seville
  - Local Institution - 0269, Valencia
- Switzerland (4):
  - Local Institution - 0291, Lausanne, Canton of Vaud
  - Local Institution - 0341, Bellinzona, Canton Ticino
  - Local Institution - 0290, Basel
  - Local Institution - 0398, Münsterlingen
- Taiwan (5):
  - Chang Gung Memorial Hospital at Kaohsiung, Kaohsiung Niao Sung Dist, Kaohsiung
  - Taipei Medical University Shuang Ho Hospital, New Taipei City
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- Turkey (Türkiye) (6):
  - Local Institution - 0361, Adana
  - Local Institution - 0365, Adana
  - Local Institution - 0383, Ankara
  - Local Institution - 0362, Ankara
  - Local Institution - 0410, Istanbul
  - Local Institution - 0364, Istanbul
- United Kingdom (11):
  - Local Institution - 0441, Exeter, Devon
  - Local Institution - 0349, Dundee, Dundee City
  - Forth Valley Royal Hospital, Larbert, Falkirk
  - Local Institution - 0189, Glasgow, Glasgow City
  - Local Institution - 0021, London, Kensington and Chelsea
  - Leicester Royal Infirmary, Leicester, Leicestershire
  - St Bartholomew's Hospital, London, London, City of
  - Local Institution - 0001, London, London, City of
  - Local Institution - 0020, Manchester
  - Local Institution - 0024, Metropolitan Borough of Wirral
  - Royal Berkshire Hospital, Reading

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT06561386.html